CLINICAL TRIAL: NCT04526587
Title: The Roswell Park Ciclib Study: A Prospective Study of Biomarkers and Clinical Features of Advanced/Metastatic Breast Cancer Treated With CDK4/6 Inhibitors
Brief Title: Biomarkers and Clinical Features of Metastatic Breast Cancer in Patients Treated With CDK4/6 Inhibitors
Status: Recruiting | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: I 571719; NCI-2020-05682 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 571719 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-08-18; First posted 2020-08-26 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue, ascites or pleural effusions, fresh body fluids or fresh biopsy,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Basic science (medical chart review, biospecimen collection): Patients electronic medical records are reviewed to capture clinical information, and patients undergo collection of blood, tissue, ascites or pleural effusions, and fresh body fluids or fresh biopsy samples for diagnosis/treatment decision, biomarker assessments, and description of mechanisms of resistance/response related to ciclib-therapy.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Diagnostic Laboratory Biomarker Analysis; Other: Medical Chart Review

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of blood, tissue, ascites or pleural effusions, and fresh body fluids or fresh biopsy samples
  Other Names: Cytologic Sampling
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Medical Chart Review — Patient's electronic health records are reviewed
  Other Names: Chart Review

SUMMARY:
This study investigates the clinical course of CDK4/6 inhibitor treated patients in the real-world setting among patients with breast cancer. CDK4/6 inhibitors may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Studying samples of blood, tissue, ascites or pleural effusions, and fresh body fluids or fresh biopsy, from patients with breast cancer that has spread to the other places in the body (metastatic) may help doctors learn more about cancer and the development of drug resistance in patients, and predict how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Delineate clinical features of disease progression and responses to subsequent therapy following progression on ciclib-based therapy.

II. Define pharmacogenomics relationships that could provide a more precise approach to drug dosing.

III. Interrogate biomarkers related to response and acquired resistance in standard clinical practice.

IV. Develop patient-derived models from resistant disease to functionally assess the mechanisms occurring with resistance.

V. Elucidate the socio-demographic features related to the use of ciclibs clinically in the Roswell Park catchment area.

OUTLINE:

Patients electronic medical records are reviewed to capture clinical information, and patients undergo collection of blood, tissue, ascites or pleural effusions, and fresh body fluids or fresh biopsy samples for diagnosis/treatment decision, biomarker assessments, and description of mechanisms of resistance/response related to ciclib-therapy.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with ER+/HER2- metastatic breast cancer or HR+/HER2-node positive, high risk early breast cancer who are being or have been treated with ciclib-based therapies are eligible for inclusion in this study

  * This includes patients receiving standard of care therapy for ER+/HER2- metastatic breast cancer, as well as those who would be eligible to participate in a non-interventional study while on a clinical study open at Roswell Park or St. Vincent's Hospital
  * Screening will occur in breast oncology clinic, by review of patient medical records for the pending, ongoing, or past treatment with ciclib-based therapy
* Participant must understand the prospective nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form

Exclusion Criteria:

* Pregnant of nursing female subjects
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with estrogen receptor positive (ER+)/HER2 negative (-) metastatic breast cancer, who are being or have been treated with ciclib-based therapies
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2030-07-03 (Estimated); Study Completion 2035-07-03 (Estimated)

PRIMARY OUTCOMES:
Collection of clinical characteristics | Up to 5 years
  Will be summarized by ciclib treatment regimen using the appropriate descriptive statistics. Differences will be evaluated using the Kruskal-Wallis and Chi-square tests, as appropriate.
Overall survival on ciclib | Up to 15 years
  Will be summarized by treatment regimen using standard Kaplan-Meier methods, with comparisons made using the log rank test. Cox regression models with time-dependent variables may be considered to account for changing treatment regimens and other patient characteristics.
Progression-free survival on ciclib | Up to 15 years
  Will be summarized by treatment regimen using standard Kaplan-Meier methods, with comparisons made using the log rank test. Cox regression models may be considered to adjust for prior therapies and other patient characteristics.
Progression-free survival on subsequent therapies | Up to 15 years
  Will be summarized by treatment regimen using standard Kaplan-Meier methods, with comparisons made using the logrank test. Cox regression models may be considered to adjust for prior therapies and other patient characteristics.
Site of the metastatic disease and time to progression | Up to 5 years
  Development of and location of metastatic disease will be summarized using the appropriate descriptive statistics.
Incidence of treatment related toxicities | Up to 5 years
  Will be summarized by ciclib treatment regimen using frequencies and relative frequencies. Comparisons may be made using Fisher's exact test. Associations between toxicity rates and patient demographic/clinical characteristics may be evaluated using logistic regression models.
Genetic variance of genes associated with ciclib metabolism | Up to 5 years
  Will be summarized in the overall sample and by treatment regimen using the appropriate descriptive statistics and graphical summaries. The association between these genetic features and toxicity and survival outcomes will be evaluated using stratified Cox regression models, where genotype will be the stratification factor. Additional models may be considered to account for other demographic or clinical characteristics. Hazard ratios with 95% confidence intervals will be obtained from model estimates.
Quantitative biomarker expressions | Up to 5 years
  Will be summarized in the overall sample and by treatment regimen using the appropriate descriptive statistics and graphical summaries. The association between baseline biomarkers and survival outcomes will be evaluated using stratified Cox regression models, where treatment regimen will be the stratification factor. Additional models may be considered to account for other demographic or clinical characteristics. Hazard ratios with 95% confidence intervals will be obtained from model estimates.
Development of patient-derived models from resistant disease | Up to 5 years
  Will be evaluated to functionally assess the mechanisms occurring with resistance. No formal statistical analyses will be performed in regards to the development of organoid and patient-derived xenograft (PDX) models.
Socio-economic features related to the use of ciclibs | Up to 5 years
  Will be elucidated clinically in the Roswell Park catchment area. Treatment regimens and sequences may be summarized by patient demographic and socio-economic characteristics using frequencies and relative frequencies. Associations may be evaluated using Chi-square tests.
Clinical course of CDK4/6 inhibitor treated patients in the "real-world" setting | Up to 5 years
  Will involve interrogating ciclib treatment patterns, treatment choices post progression, toxicities, clinical responses following progression, and ultimately differences in overall survival.

OTHER OUTCOMES:
Examination of biomarkers of response | Up to 5 years
  Will examine biomarkers of response/resistance and association with long term outcomes relative to pretreatment controls.
Single-nucleotide polymorphisms | Day 8 to day 18 of cycle 1
  Blood will be collected to interrogate single-nucleotide polymorphisms in CYP3A4 and related genes associated with metabolism of ciclib compounds. These polymorphisms will be related to dose limiting toxicities and dose interruptions. Blood samples for pharmacokinetic and pharmacogenomic analysis will be drawn during regular laboratory blood draws.
Circulating cell free DNA (cfDNA) | Up to 5 years
  Serial peripheral blood samples will be prospectively collected at specified time points and processed for cfDNA and circulating tumor cells (CTC) isolation. CTCs will be utilized for the development of 3-dimensional (3D) organoid cultures and CTC-derived xenograft models.
Development of functional models (patient-derived models) from individuals with progressive disease | Up to 5 years
  Will only employ tissues and /or body fluids that are being discarded or do not involve any additional procedures for the patients. This includes, excess tissue that is not required for diagnosis or pleural effusions or peritoneal ascites. Cells isolated from the samples will be used for the development of organoid or PDX models.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka K Witkiewicz, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] O'Connor TN, Schultz E, Kabraji S, Levine E, Williams AJ, Knudsen ES, Witkiewicz AK. Real-World Plasma Thymidine Kinase Activity in High-Risk and Metastatic Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Breast Cancer Treated With Cyclin-Dependent Kinase 4/6 Inhibitors. JCO Precis Oncol. 2026 Jan;10:e2500346. doi: 10.1200/PO-25-00346. Epub 2026 Jan 23. PMID 41576303
- [Derived] Tzetzo SL, Schultz E, Wang J, Rosenheck HR, Mahan S, Knudsen ES, Witkiewicz AK. Baseline cell cycle and immune profiles indicate CDK4/6 inhibitor response in metastatic HR + /HER2- breast cancer. NPJ Breast Cancer. 2025 Jun 12;11(1):54. doi: 10.1038/s41523-025-00767-2. PMID 40506447
- [Derived] Witkiewicz AK, Schultz E, Wang J, Hamilton D, Levine E, O'Connor T, Knudsen ES. Determinants of response to CDK4/6 inhibitors in the real-world setting. NPJ Precis Oncol. 2023 Sep 13;7(1):90. doi: 10.1038/s41698-023-00438-0. PMID 37704753